CLINICAL TRIAL: NCT06320093
Title: Training Social and Health Care prOfessionals in mUsic-based Therapeutic iNterventions to Support Older People With Dementia
Acronym: SOUND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_002_2024
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Dementia; Older People
Keywords: dementia; older people; music; caregiver
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sound intervention (Experimental): the SOUND intervention is a new and innovative method of applying musical activities in a circle consisting of elderly people with mild-to-moderate dementia, caregivers, family caregivers and young people.
  Interventions: Other: SOUND Intervention

INTERVENTIONS:
Other: SOUND Intervention — The intervention involved active (vocal and rhythmic production) and passive (listening to musical pieces) musical activities accompanied by motor coordination exercises. It consisted of 12 meetings (2 per week for 6 weeks) of 45 minutes each.

SUMMARY:
The study will investigate the effects of an inovative intervention based on the use of music on 45 professionals in the field of dementia, 45 elderly people with dementia.

DETAILED DESCRIPTION:
The study aims to develop an innovative therapeutic intervention (SOUND intervention) based on the use of music to improve behavior, mood, well-being, and maintain cognitive function in older people with dementia.

The study will investigate the effects of the SOUND intervention on 45 professionals in the field of dementia, 45 elderly people with dementia, and 5 family caregivers by monitoring quantitative outcome variables that will be measured through psychometric and qualitative scales interpreted through open-ended questions and observations.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate dementia
* no severe hearing and visual impairment or motor problems

Exclusion Criteria:

* no formal caregiver
* no informal caregiver

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in mental wellbeing of patients with dementia | baseline, 12 and 14 weeks later
  The World Health Organisation- Five Well-Being Index (WHO-5) is a short self-reported measure of current mental wellbeing.The WHO-5 consists of five statements, which respondents rate according to the scale below (in relation to the past two weeks): All of the time = 5; Most of the time = 4; More than half of the time = 3; Less than half of the time = 2 Some of the time = 1; At no time = 0. The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Change in cognitive status of patients with dementia | baseline, 12 and 14 weeks later
  The cognitive status has been evaluated by the Montreal Cognitive Assessment (MOCA) test. MOCA is an assessment tool used globally to detect early onset of dementia among people of old age. The tool is a one-page 30-point test that the physician can administer to check the memory, language, recall, and other markers of cognitive acuity of a patient. Normal cognition: 26-30 points; Mild Cognitive Impairment: 18-25 points; Moderate Cognitive Impairment: 10-17 points; Severe Cognitive Impairment: under 10 points.
Change in stress of health care providers | baseline, 12 and 14 weeks later
  The Burnout Assessment Tool (BAT) is a self-assessment questionnaire that measures parameters associated with Burnout. All items are expressed as statements with five frequency-based response categories (1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always). The total burnout score is calculated as a mean of all 23 items, and a high score is indicative of high levels of burnout.

CONTACTS AND LOCATIONS:
Locations (3):
- INRCA Hospital, Ancona, Italy
- Sons do Estamine Associacao, Trofa, Portugal
- Associatia Habilitas, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No